CLINICAL TRIAL: NCT04475848
Title: A Randomized, Investigator- /Subject-blind, Single- and Multiple-ascending Dose, Placebo-controlled Study to Investigate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of RO6953958 (Including RO6953958 Effect on Midazolam) Following Oral Administration in Healthy Male Participants
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of RO6953958 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP41695; 2019-004486-41 (EudraCT Number)
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Autistic Disorder; Autism Spectrum Disorder; Child Development Disorders, Pervasive; Mental Disorders; Neurodevelopmental Disorders
Keywords: Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Child Development Disorders, Pervasive; Mental Disorders; Neurodevelopmental Disorders | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1: SAD/FE (Experimental): There will be 7 cohorts in this study. In each cohort, participants will receive a single oral dose of RO6953958 while fasted. Participants in the fed (FE) cohort will return to receive the same single oral dose of RO6953958 repeated in the fed state.
  Interventions: Drug: RO6953958
- Part 1: SAD placebo (Placebo Comparator): There will be 7 cohorts in this study. In each cohort, participants will receive a single oral dose of a placebo while fasted/fed.
  Interventions: Drug: Placebo
- Part 2: MAD (Experimental): A maximum of 5 dose levels are anticipated. For each dose level, a minimum of 8 and a maximum of 16 participants will receive a multiple oral dose of RO6953958 once daily (QD) for 10 days.
  Interventions: Drug: RO6953958
- Part 2: MAD placebo (Placebo Comparator): A maximum of 5 dose levels are anticipated. For each dose level, a minimum of 8 and a maximum of 16 participants will receive a multiple oral dose of palcebo QD for 10 days.
  Interventions: Drug: Placebo
- Part 3: DDI (Experimental): RO6953958 will be administered at the maximum dose QD that was tested in the ongoing Part 2 (MAD).
  Participants will also be administered midazolam.
  Interventions: Drug: RO6953958; Drug: Midazolam

INTERVENTIONS:
Drug: RO6953958 — Part 1: RO6953958 will be administered in an adaptive manner. The starting dose is planned to be 5 milligrams (mg).
  Part 2: The starting dose is planned to be 45 mg.
  Part 3: RO6953958 will be administered QD following a standardized breakfast on Day 3 to Day 14 at the maximum dose QD that was tested in the ongoing Part 2 (MAD).
  Arms: Part 1: SAD/FE; Part 2: MAD; Part 3: DDI
Drug: Placebo — Part 1: A placebo will be administered in an adaptive manner. The starting dose is planned to be 5 mg.
  Part 2: The starting dose is planned to be 45 mg.
  Arms: Part 1: SAD placebo; Part 2: MAD placebo
Drug: Midazolam — Midazolam will be administered as single intervenous (IV) bolus injection of 100 micrograms (ug) on Day 1 and Day 13, and as single oral dose of 300 ug on Day 2 and Day 14.
  Arms: Part 3: DDI

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single- and multiple-ascending doses (SAD (Part 1) and MAD (Part 2)) and food effect (FE) of RO6953958 following oral administration in healthy male participants. Part 3 (Drug-drug interaction (DDI)) will assess the safety, tolerability, and effect of RO6953958 on the PK of the cytochrome P450 (CYP) 3A substrate midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) within 18 to 31 kg/m2
* During treatment and for at least 14 days after the last dose to remain abstinent
* Refrain from donating sperm for at least 14 days after last dose
* Part 2 (MAD) only - Participants must be prepared to collect a sleep log and wear an actigraphy device the week before participation in the study. Participants must also have scored 5 or less on the Pittsburgh Sleep Quality Index (PSQI), less than 13 on the Epworth sleepiness scale (ESS), and not be considered an extreme morning or evening type according to the morningness-eveningness questionnaire (MEQ) at screening to be eligible.

Exclusion Criteria:

* History or evidence of any medical condition potentially altering the absorption, metabolism, or elimination of drugs
* History of any clinically significant gastrointestinal, renal, hepatic, bronchopulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological, or allergic disease, sleep disorders (Part 2 [MAD] only), unexplained syncope (within 12 months prior to screening), metabolic disorder, cancer, or cirrhosis
* Use of any psychoactive medication, or medications known to have effects on central nervous system (CNS), or blood flow
* History of convulsions
* History of clinically significant hypersensitivity (e.g., drugs, excipients) or allergic reactions
* Abnormal blood pressure (BP) and pulse rate
* Presence of orthostatic hypotension
* History or presence of clinically significant ECG abnormalities or cardiovascular disease
* Current or chronic history of liver disease or known hepatic or biliary abnormalities
* Known active or any major episode of infection within 4 weeks prior to the start of drug administration
* Participants who test positive for acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
* Have used or intend to use over-the-counter (OTC) or prescription medication including herbal medications within 30 days prior to dosing
* Positive test for drugs, abuse of alcohol, human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus (HCV), presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test
* Inability or unwillingness to fully consume standardized breakfast at Day 1
* Part 2 (MAD) only - Participants who have issues sleeping or participants who have travelled across 2 or more time zones in the past month.
* Part 2 (MAD) only - Participants who cannot produce sufficient saliva for study assessments
* Participants who have donated more than 500 mL of blood or blood products or had significant blood loss within 3 months prior to screening
* Have a history of clinically significant back pain, back pathology, and/or back injury that may predispose to complications from, or technical difficulty with, lumbar puncture
* Complications that would lead to difficulty in obtaining a lumbar puncture
* Part 3 (DDI) only - History of hypersensitivity to benzodiazepines (including midazolam) or its formulation ingredients

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 88 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Hammersmith Medicines Research; Central Middlesex Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one centre in the United Kingdom.
Groups:
- Part 1 (SAD): RO6953958 5mg (Fasted); Part 1 (SAD): RO6953958 15mg (Fasted); Part 1 (SAD): RO6953958 45mg (Fasted); Part 1 (SAD): RO6953958 180mg (Fasted); Part 1 (SAD): RO6953958 360mg (Fasted): Participants received a single oral dose of RO6953958 while fasted.
- Part 1 (SAD): RO6953958 90mg (Fasted or Fed): Participants received a single oral dose of RO6953958 while fasted. Participants in the fed (FE) cohort returned to receive the same single oral dose of RO6953958 repeated in the fed state.
- Part 1 (SAD): Placebo (Fasted): Participants received a single oral dose of a placebo while fasted.
- Part 1 (SAD): Placebo (Fed): Participants received a single oral dose of a placebo while fed.
- Part 2 (MAD): RO6953958 45mg: Participants received a multiple oral dose of RO6953958 once daily (QD) for 10 days.
- Part 2 (MAD): RO6953958 140mg; Part 2 (MAD): RO6953958 210mg: Participants received a multiple oral dose of RO6953958 QD for 10 days.
- Part 2 (MAD): Placebo: Participants received a multiple oral dose of a placebo QD for 10 days.
- Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug: Participants were administered RO6953958 at the maximum dose QD that was tested in the ongoing Part 2 (MAD). Participants were also administered midazolam.
Period: Overall Study
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted or Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 1 (SAD): Placebo (Fasted) | Part 1 (SAD): Placebo (Fed) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 2 (MAD): Placebo | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Started | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 6 | 6 | 6 | 6 | 16
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 6 | 6 | 6 | 6 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted or Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 1 (SAD): Placebo (Fasted) | Part 1 (SAD): Placebo (Fed) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 2 (MAD): Placebo | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 6 | 6 | 6 | 6 | 16 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (9.9) | 37.3 (8.1) | 37.5 (4.3) | 33.7 (11.9) | 40.3 (10.3) | 33.8 (12.6) | 34.1 (9.7) | 38.5 (2.1) | 32.5 (7.4) | 36.2 (11.7) | 38.7 (12.9) | 30.3 (11.2) | 33.6 (10.6) | 35.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 6 | 6 | 6 | 6 | 16 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 5 | 5 | 5 | 6 | 6 | 5 | 9 | 2 | 6 | 6 | 6 | 6 | 16 | 83
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 8
  White | 3 | 3 | 5 | 6 | 5 | 6 | 9 | 2 | 6 | 4 | 2 | 4 | 10 | 65
  More than one race | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Parts 1, 2 and 3: Percentage of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Part 1: From randomization up to 7 weeks (or up to 14 weeks if the participant is part of the food effect cohort). Parts 2 and 3: From randomization up to 8 weeks
Population: The safety population included all participants randomized to study treatment and who received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted or Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 1 (SAD): Placebo (Fasted) | Part 1 (SAD): Placebo (Fed) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 2 (MAD): Placebo | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 6 | 6 | 6 | 6 | 16
Participants | 2 | 2 | 2 | 4 | 2 | 3 | 2 | 0 | 4 | 6 | 4 | 2 | 15

2. Primary Outcome: Part 2: Number of Participants With Post-baseline Suicide Risk, Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a questionnaire that is used to assess a participant's suicidal ideation and behaviors. The categories in the questionnaire have binary responses (yes/no) and include: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation or behavior is indicated by a "yes" answer to any of the listed categories. A score of 0 is assigned if no suicide risk is present. Categories with non-zero values are reported here.
Time Frame: From randomization up to 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Suicidal Ideation or Behavior | 0 | 0 | 0 | 0
  Highest Suicidal Behavior | 0 | 0 | 0 | 0
  Highest Suicidal Ideation | 0 | 0 | 0 | 0
  Self-Injury Behavior w/o suicidal intent | 0 | 0 | 0 | 0

3. Secondary Outcome: Parts 1, 2 and 3: Maximum Observed Plasma Concentration (Cmax) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The pharmacokinetic (PK) population included all participants who received active (RO6953958) treatment.
Measure: Mean (Standard Deviation); unit: Nanograms per Milliliter (ng/mL)
Groups:
- Part 1 (SAD): RO6953958 90mg (Fasted); Part 1 (SAD): RO6953958 180mg (Fasted); Part 1 (SAD): RO6953958 360mg (Fasted): Participants received a single oral dose of RO6953958 while fasted.
- Part 1 (SAD): RO6953958 90mg (Fed): Participants in the fed (FE) cohort returned to receive the same single oral dose of RO6953958 repeated in the fed state.
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Nanograms per Milliliter (ng/mL)
  RO6953958 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
  RO6953958 - Day 1 | 70.3 (31.4) | 150 (34.2) | 299 (50.0) | 451 (30.7) | 932 (34.6) | 618 (47.4) | 866 (39.5) | 490 (25.0) | 1250 (49.7) | 1580 (21.8) |
  RO6953958 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO6953958 - Day 3 |  |  |  |  |  |  |  |  |  |  | 1850 (30.5)
  RO6953958 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO6953958 - Day 10 |  |  |  |  |  |  |  | 490 (25.0) | 1250 (49.7) | 1580 (21.8) |
  RO6953958 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO6953958 - Day 14 |  |  |  |  |  |  |  |  |  |  | 2120 (32.8)
  RO7021594 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
  RO7021594 - Day 1 | 61.3 (45.0) | 187 (41.0) | 480 (76.0) | 490 (18.8) | 819 (21.2) | 1230 (67.2) | 3.57 (28.3) | 1850 (21.6) | 677 (47.9) | 1100 (41.4) |
  RO7021594 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7021594 - Day 3 |  |  |  |  |  |  |  |  |  |  | 2890 (61.9)
  RO7021594 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO7021594 - Day 10 |  |  |  |  |  |  |  | 1100 (41.4) | 3180 (76.7) | 6010 (65.3) |
  RO7021594 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7021594 - Day 14 |  |  |  |  |  |  |  |  |  |  | 5310 (66.7)
  RO7045755 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
  RO7045755 - Day 1 | 32.3 (29.6) | 77.3 (25.2) | 169 (36.9) | 272 (32.5) | 491 (29.1) | 1.69 (71.1) | 1.33 (42.4) | 171 (43.0) | 452 (31.5) | 629 (30.3) |
  RO7045755 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7045755 - Day 3 |  |  |  |  |  |  |  |  |  |  | 710 (34.9)
  RO7045755 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO7045755 - Day 10 |  |  |  |  |  |  |  | 194 (44.9) | 456 (68.3) | 528 (46.7) |
  RO7045755 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7045755 - Day 14 |  |  |  |  |  |  |  |  |  |  | 816 (42.1)

4. Secondary Outcome: Parts 2 and 3: Average Plasma Concentration (Cavg) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The pharmacokinetic (PK) population included all participants who received active (RO6953958) treatment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 16
ng/mL
  RO6953958 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO6953958 - Day 1 | 81.47 (28.35) | 279.87 (163.45) | 496.48 (128.30) |
  RO6953958 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO6953958 - Day 3 |  |  |  | 531.60 (276.14)
  RO6953958 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO6953958 - Day 10 | 87.96 (26.59) | 283.22 (141.49) | 410.99 (161.04) |
  RO6953958 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO6953958 - Day 14 |  |  |  | 646.81 (453.67)
  RO7021594 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7021594 - Day 1 | 407.07 (185.06) | 1380.91 (931.78) | 2987.02 (1307.84) |
  RO7021594 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7021594 - Day 3 |  |  |  | 2305.32 (1570.98)
  RO7021594 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7021594 - Day 10 | 743.87 (336.40) | 2759.37 (2433.54) | 4822.34 (2550.00) |
  RO7021594 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7021594 - Day 14 |  |  |  | 4552.31 (3813.18)
  RO7045755 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7045755 - Day 1 | 69.97 (33.67) | 194.92 (116.77) | 293.36 (146.13) |
  RO7045755 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7045755 - Day 3 |  |  |  | 341.71 (165.07)
  RO7045755 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7045755 - Day 10 | 76.29 (38.08) | 230.74 (169.20) | 272.07 (204.45) |
  RO7045755 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7045755 - Day 14 |  |  |  | 428.80 (303.11)

5. Secondary Outcome: Parts 1, 2 and 3: Time to Reach Maximum Observed Plasma Concentration (Tmax) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The pharmacokinetic (PK) population included all participants who received active (RO6953958) treatment.
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Hours (h)
  RO6953958 - Day 1 | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 2.12] | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 2.02] | 4.00 [2.00 to 5.00] | 2.00 [1.00 to 5.00] | 2.00 [0.50 to 3.00] | 2.53 [2.00 to 3.00] | 2.01 [1.00 to 3.02] | 3.00 [2.00 to 3.02] | 3.00 [2.00 to 5.08]
  RO6953958 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO6953958 - Day 3 |  |  |  |  |  |  |  |  |  |  | 3.00 [2.00 to 5.08]
  RO6953958 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO6953958 - Day 10 |  |  |  |  |  |  |  | 2.02 [1.00 to 3.00] | 2.04 [1.02 to 3.00] | 2.00 [1.00 to 3.00] |
  RO6953958 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO6953958 - Day 14 |  |  |  |  |  |  |  |  |  |  | 3.00 [2.00 to 5.00]
  RO7021594 - Day 1 | 2.00 [1.00 to 3.00] | 2.00 [2.00 to 6.00] | 5.50 [5.00 to 7.00] | 6.51 [5.00 to 10.00] | 5.50 [3.00 to 10.00] | 6.50 [2.00 to 48.02] | 7.01 [5.00 to 24.05] | 5.00 [3.00 to 6.03] | 3.02 [3.00 to 10.00] | 5.00 [3.00 to 7.00] | 6.02 [3.00 to 10.08]
  RO7021594 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7021594 - Day 3 |  |  |  |  |  |  |  |  |  |  | 5.08 [3.00 to 12.00]
  RO7021594 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO7021594 - Day 10 |  |  |  |  |  |  |  | 5.02 [2.08 to 5.05] | 4.00 [3.00 to 7.00] | 4.01 [3.00 to 7.03] |
  RO7021594 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7021594 - Day 14 |  |  |  |  |  |  |  |  |  |  | 6.02 [3.00 to 10.08]
  RO7045755 - Day 1 | 1.50 [1.00 to 3.00] | 2.00 [1.00 to 6.00] | 4.00 [2.02 to 6.00] | 5.00 [3.00 to 6.00] | 5.00 [2.00 to 7.00] | 4.00 [2.00 to 7.05] | 5.01 [3.00 to 10.00] | 4.00 [3.00 to 5.00] | 3.02 [3.00 to 5.00] | 4.08 [2.00 to 6.02] | 5.00 [3.00 to 10.03]
  RO7045755 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7045755 - Day 3 |  |  |  |  |  |  |  |  |  |  | 4.02 [2.05 to 6.02]
  RO7045755 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO7045755 - Day 10 |  |  |  |  |  |  |  | 3.01 [2.08 to 5.02] | 3.04 [3.00 to 5.00] | 2.51 [2.00 to 6.03] |
  RO7045755 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7045755 - Day 14 |  |  |  |  |  |  |  |  |  |  | 5.00 [3.00 to 10.03]

6. Secondary Outcome: Part 1: Last Quantifiable Concentration (Clast) of RO6953958 and Its Metabolites RO7021594 and RO7045755 in Fasted and Fed State
Time Frame: Day 1-10
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 1 (SAD): Placebo (Fasted) | Part 1 (SAD): Placebo (Fed)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0
ng/mL
  RO6953958 | 3.88 (63.7) | 4.42 (71.6) | 5.98 (82.4) | 6.75 (98.2) | 11.1 (130.4) | 8.99 (97.7) | 10.6 (67.1) |  |
  RO7021594 | 2.67 (24.0) | 6.22 (84.1) | 12.6 (163.1) | 41.1 (3.16) | 31.6 (4.04) | 80.3 (12.6) | 115.1 (9.75) |  |
  RO7045755 | 5.64 (53.3) | 7.48 (55.7) | 6.52 (78.2) | 84.4 (7.71) | 116.6 (6.70) | 59.3 (6.15) | 60.7 (6.25) |  |

7. Secondary Outcome: Part 1: Time To the Last Quantifiable Concentration (Tlast) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-10
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h
  RO6953958 | 9.44 (25.0) | 16.47 (43.8) | 21.40 (28.9) | 51.37 (16.6) | 24.00 (0.0) | 70.14 (22.3) | 88.77 (32.1)
  RO7021594 | 87.23 (14.9) | 96.03 (0.1) | 96.01 (0.0) | 170.15 (29.3) | 144.29 (24.6) | 208.08 (10.8) | 216.78 (0.5)
  RO7045755 | 3.84 (52.9) | 19.06 (37.0) | 26.96 (28.9) | 54.96 (21.2) | 38.10 (37.0) | 74.87 (12.2) | 92.34 (34.9)

8. Secondary Outcome: Parts 1, 2 and 3: Terminal Elimination Phase Half-Life (t1/2) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
h
  RO6953958 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 3 | 0
  RO6953958 - Day 1 | 1.75 (11.8) | 3.43 (52.4) | 3.98 (46.3) | 9.54 (13.9) | 3.57 (20.6) | 13.1 (23.7) | 14.9 (21.8) | 2.63 (43.6) | 6.60 (18.9) | 4.99 (27.3) |
  RO6953958 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14
  RO6953958 - Day 3 |  |  |  |  |  |  |  |  |  |  | 5.87 (27.6)
  RO6953958 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 3 | 0
  RO6953958 - Day 10 |  |  |  |  |  |  |  | 3.43 (42.7) | 7.90 (51.0) | 6.29 (15.6) |
  RO6953958 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO6953958 - Day 14 |  |  |  |  |  |  |  |  |  |  | 6.20 (56.2)
  RO7021594 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
  RO7021594 - Day 1 | 21.0 (13.7) | 19.7 (12.4) | 19.1 (14.1) | 20.8 (25.4) | 20.6 (30.4) | 27.7 (18.6) | 27.1 (17.3) |  |  |  |
  RO7021594 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RO7021594 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO7021594 - Day 10 |  |  |  |  |  |  |  | 31.5 (31.2) | 34.0 (9.7) | 35.8 (17.5) |
  RO7021594 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7021594 - Day 14 |  |  |  |  |  |  |  |  |  |  | 36.0 (24.9)
  RO7045755 - Day 1: number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 0
  RO7045755 - Day 1 | 3.84 (52.9) | 4.54 (31.9) | 4.82 (26.0) | 10.3 (15.7) | 5.25 (13.1) | 13.5 (22.8) | 12.7 (20.6) | 3.89 (42.9) | 5.38 (33.6) | 6.21 (15.2) |
  RO7045755 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14
  RO7045755 - Day 3 |  |  |  |  |  |  |  |  |  |  | 5.33 (28.0)
  RO7045755 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 4 | 0
  RO7045755 - Day 10 |  |  |  |  |  |  |  | 4.39 (50.6) | 6.72 (42.9) | 7.91 (54.4) |
  RO7045755 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7045755 - Day 14 |  |  |  |  |  |  |  |  |  |  | 5.81 (55.8)

9. Secondary Outcome: Parts 2 and 3: Area Under the Concentration-Time Curve (AUC(0-t)) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 16
h*ng/mL
  RO6953958 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO6953958 - Day 1 | 1830 (44.7) | 5820 (63.9) | 11600 (27.5) |
  RO6953958 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO6953958 - Day 3 |  |  |  | 11400 (51.2)
  RO6953958 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO6953958 - Day 10 | 2010 (38.4) | 6060 (58.0) | 9180 (44.9) |
  RO6953958 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO6953958 - Day 14 |  |  |  | 14300 (65.1)
  RO7021594 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7021594 - Day 1 | 9040 (43.8) | 27400 (79.8) | 64000 (62.0) |
  RO7021594 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7021594 - Day 3 |  |  |  | 47000 (60.0)
  RO7021594 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7021594 - Day 10 | 16400 (47.9) | 51500 (85.4) | 103000 (59.3) |
  RO7021594 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7021594 - Day 14 |  |  |  | 153000 (82.6)
  RO7045755 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7045755 - Day 1 | 1450 (74.0) | 3980 (70.8) | 6290 (56.5) |
  RO7045755 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7045755 - Day 3 |  |  |  | 7240 (57.7)
  RO7045755 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7045755 - Day 10 | 1550 (79.6) | 4290 (97.2) | 5120 (88.8) |
  RO7045755 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7045755 - Day 14 |  |  |  | 9560 (86.4)

10. Secondary Outcome: Part 1: Area Under the Plasma Concentration Versus Time Curve From Zero to 24h Postdose (AUC(0-24h)) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-5
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL
  RO6953958 | 204 (38.9) | 665 (51.3) | 1740 (26.8) | 4140 (39.9) | 5330 (38.9) | 6170 (39.7) | 8720 (70.9)
  RO7021594 | 829 (38.4) | 2910 (45.1) | 7410 (81.6) | 9010 (17.9) | 12500 (24.7) | 22700 (60.9) | 23100 (28.9)
  RO7045755 | 238 (53.2) | 707 (45.3) | 1610 (34.7) | 3870 (28.3) | 5330 (31.1) | 4340 (70.4) | 6630 (68.5)

11. Secondary Outcome: Part 1: Area Under the Plasma Concentration Versus Time Curve From Zero to the Last Measurable Concentration (AUC0-last) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-10
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL
  RO6953958 | 188 (38.7) | 651 (52.4) | 1730 (27.7) | 4990 (46.1) | 5330 (38.9) | 9470 (31.6) | 14700 (83.0)
  RO7021594 | 1410 (38.6) | 4940 (48.7) | 12200 (89.0) | 21000 (42.0) | 21400 (40.1) | 74000 (79.2) | 78500 (46.2)
  RO7045755 | 208 (56.0) | 684 (50.5) | 1650 (34.6) | 4970 (32.3) | 5670 (34.0) | 6740 (63.6) | 11500 (93.0)

12. Secondary Outcome: Part 1: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-10
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL
  RO6953958 | 206 (39.7) | 676 (52.2) | 1780 (26.2) | 5120 (46.5) | 5410 (39.3) | 9710 (31.3) | 15200 (78.7)
  RO7021594 | 1190 (36.8) | 4160 (46.5) | 10500 (85.3) | 15300 (28.3) | 18100 (33.3) | 44800 (68.5) | 45400 (30.3)
  RO7045755 | 249 (57.3) | 738 (48.8) | 1700 (35.4) | 4880 (31.3) | 5750 (33.1) | 6140 (65.8) | 9680 (79.3)

13. Secondary Outcome: Parts 1, 2 and 3: Apparent Clearance (CL/F) of RO6953958
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
L/h
  Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 0
  Day 1 | 24.3 (39.7) | 22.2 (52.2) | 25.2 (26.2) | 17.6 (46.5) | 16.6 (39.3) | 18.5 (31.3) | 23.7 (78.7) | 24.6 (44.7) | 22.0 (66.7) | 17.2 (26.4) |
  Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  Day 3 |  |  |  |  |  |  |  |  |  |  | 18.43 (51.2)
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 3 | 0
  Day 10 |  |  |  |  |  |  |  | 22.4 (38.4) | 23.1 (58.0) | 17.4 (27.8) |
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  Day 14 |  |  |  |  |  |  |  |  |  |  | 15.87 (58.6)

14. Secondary Outcome: Parts 1, 2 and 3: Apparent Volume of Distribution (V/F) of RO6953958
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
L
  Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
  Day 1 | 89.1 (51.2) | 110 (47.5) | 145 (42.7) | 242 (45.3) | 85.8 (35.8) | 45.5 (425) | 509 (91.5) | 93.1 (30.2) | 209 (63.0) | 164 (69.6) |
  Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  Day 3 |  |  |  |  |  |  |  |  |  |  | 161 (58.3)
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 3 | 0
  Day 10 |  |  |  |  |  |  |  | 111 (25.2) | 263 (77.2) | 158 (42.1) |
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  Day 14 |  |  |  |  |  |  |  |  |  |  | 142 (72.5)

15. Secondary Outcome: Parts 1 and 2: Cumulative Amount of Unchanged Drug Excreted Into the Urine (Ae) of RO6953958
Time Frame: Day 1 and 10
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mg
  Day 1 | 0.0322 (0.00658) | 0.133 (0.0513) | 0.266 (0.0766) | 0.612 (0.245) | 0.321 (0.0831) | 0.675 (0.377) | 1.14 (0.465) | 0.192 (0.0814) | 0.525 (0.234) | 0.461 (0.203)
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 6
  Day 10 |  |  |  |  |  |  |  | 0.220 (0.111) | 0.562 (0.260) | 0.437 (0.311)

16. Secondary Outcome: Parts 1 and 2: Fraction of the Administered Drug Excreted Into the Urine (Fe) of RO6953958
Time Frame: Day 1 and 10
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mg
  Day 1 | 0.644 (0.132) | 0.888 (0.342) | 0.592 (0.170) | 0.679 (0.272) | 0.356 (0.0923) | 0.375 (0.209) | 0.316 (0.129) | 0.426 (0.181) | 0.375 (0.167) | 0.220 (0.0965)
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 6
  Day 10 |  |  |  |  |  |  |  | 0.490 (0.246) | 0.402 (0.186) | 0.208 (0.148)

17. Secondary Outcome: Parts 1 and 2: Renal Clearance of the Drug From Urine (CLR) of RO6953958
Time Frame: Day 1 and 10
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
mg
  Day 1 | 115 (139.3) | 142 (52.8) | 123 (65.9) | 116 (59.6) | 49.9 (60.7) | 56.2 (150.2) | 81.7 (66.0) | 97.3 (29.5) | 84.3 (50.7) | 36.5 (35.3)
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6
  Day 10 |  |  |  |  |  |  |  | 91.4 (43.5) | 78.7 (51.0) | 37.3 (36.3)

18. Secondary Outcome: Parts 2 and 3: Trough Plasma Concentration (Ctrough) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1, 3, 10, 12, 13
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 16
ng/mL
  RO6953958 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO6953958 - Day 1 | 0.473 (1305.9) | 31.0 (160.4) | 82.4 (50.2) |
  RO6953958 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO6953958 - Day 3 |  |  |  | 60.78 (116.9)
  RO6953958 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO6953958 - Day 10 | 1.20 (660.9) | 24.2 (177.7) | 40.5 (161.4) |
  RO6953958 - Day 12: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO6953958 - Day 12 |  |  |  | 57.89 (190.9)
  RO6953958 - Day 13: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO6953958 - Day 13 |  |  |  | 54.40 (197.6)
  RO7021594 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7021594 - Day 1 | 227 (48.0) | 704 (99.0) | 2130 (60.4) |
  RO7021594 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7021594 - Day 3 |  |  |  | 1462.36 (67.3)
  RO7021594 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7021594 - Day 10 | 449 (52.2) | 1390 (98.8) | 3020 (62.9) |
  RO7021594 - Day 12: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7021594 - Day 12 |  |  |  | 2566.84 (95.0)
  RO7021594 - Day 13: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7021594 - Day 13 |  |  |  | 2517.91 (86.1)
  RO7045755 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7045755 - Day 1 | 4.25 (930.3) | 27.6 (300.4) | 63.0 (119.7) |
  RO7045755 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7045755 - Day 3 |  |  |  | 62.88 (199.9)
  RO7045755 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7045755 - Day 10 | 5.14 (1196.9) | 33.6 (232.9) | 31.7 (429.6) |
  RO7045755 - Day 12: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7045755 - Day 12 |  |  |  | 73.42 (283.5)
  RO7045755 - Day 13: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7045755 - Day 13 |  |  |  | 63.54 (276.8)

19. Secondary Outcome: Parts 2 and 3: Accumulation Ratio Based on AUC (RAUC) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 16
Ratio of AUC
  RO6953958 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO6953958 - Day 10 | 1.10 (8.4) | 1.04 (15.9) | 0.794 (23.9) |
  RO6953958 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO6953958 - Day 14 |  |  |  | 1.25 (24.4)
  RO7021594 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7021594 - Day 10 | 1.81 (13.9) | 1.87 (22.3) | 1.60 (21.8) |
  RO7021594 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7021594 - Day 14 |  |  |  | 3.27 (52.6)
  RO7045755 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7045755 - Day 10 | 1.07 (8.1) | 1.08 (23.4) | 0.814 (31.2) |
  RO7045755 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7045755 - Day 14 |  |  |  | 1.32 (35.8)

20. Secondary Outcome: Parts 2 and 3: Accumulation Ratio Based on Cmax (RCmax) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of Cmax
Arm/Group | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 16
Ratio of Cmax
  RO6953958 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO6953958 - Day 10 | 1.05 (19.0) | 1.05 (24.0) | 0.856 (13.6) |
  RO6953958 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO6953958 - Day 14 |  |  |  | 1.14 (27.0)
  RO7021594 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7021594 - Day 10 | 1.63 (12.1) | 1.77 (32.2) | 1.59 (16.8) |
  RO7021594 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7021594 - Day 14 |  |  |  | 1.84 (38.2)
  RO7045755 - Day 10: number analyzed (Participants) | 6 | 6 | 6 | 0
  RO7045755 - Day 10 | 1.13 (10.0) | 1.01 (45.2) | 0.839 (28.1) |
  RO7045755 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 16
  RO7045755 - Day 14 |  |  |  | 1.15 (30.6)

21. Secondary Outcome: Parts 2 and 3: Accumulation Ratio Based on Ctrough (RCtrough) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment. No data were analyzed and this outcome measure was not conducted.
Arm/Group | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Parts 1, 2 and 3: Molecular Weight Adjusted Metabolite-to-Parent Ratio for Cmax of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Metabolite Ratio for Cmax
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Metabolite Ratio for Cmax
  RO7021594 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
  RO7021594 - Day 1 | 0.839 (61.6) | 1.20 (43.3) | 1.54 (42.3) | 1.05 (32.1) | 0.846 (37.2) | 1.91 (85.3) | 1.43 (43.4) | 1.39 (77.7) | 1.45 (99.3) | 1.97 (72.9) |
  RO7021594 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7021594 - Day 3 |  |  |  |  |  |  |  |  |  |  | 1.50 (72.4)
  RO7021594 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO7021594 - Day 10 |  |  |  |  |  |  |  | 2.16 (50.7) | 2.46 (109.8) | 3.66 (69.0) |
  RO7021594 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7021594 - Day 14 |  |  |  |  |  |  |  |  |  |  | 2.41 (62.8)
  RO7045755 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
  RO7045755 - Day 1 | 0.442 (16.9) | 0.497 (29.5) | 0.544 (37.9) | 0.580 (24.7) | 0.507 (17.6) | 0.474 (38.0) | 0.534 (40.3) | 0.350 (32.3) | 0.366 (35.6) | 0.328 (27.2) |
  RO7045755 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7045755 - Day 3 |  |  |  |  |  |  |  |  |  |  | 0.369 (24.8)
  RO7045755 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO7045755 - Day 10 |  |  |  |  |  |  |  | 0.380 (37.3) | 0.352 (29.4) | 0.321 (38.1) |
  RO7045755 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7045755 - Day 14 |  |  |  |  |  |  |  |  |  |  | 0.371 (33.9)

23. Secondary Outcome: Parts 1, 2 and 3: Molecular Weight Adjusted Metabolite-to-Parent Ratio for Area Under the Concentration-Time Curve (AUC(0-t)) of RO6953958 and Its Metabolites RO7021594 and RO7045755
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Metabolite Ratio for AUC(0-t)
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Metabolite Ratio for AUC(0-t)
  RO7021594 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
  RO7021594 - Day 1 | 6.98 (73.9) | 7.30 (48.6) | 6.81 (69.3) | 3.97 (34.0) | 3.84 (32.6) | 7.39 (68.6) | 5.02 (50.3) | 4.75 (72.5) | 5.31 (90.8) | 5.32 (77.9) |
  RO7021594 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7021594 - Day 3 |  |  |  |  |  |  |  |  |  |  | 0.612 (40.0)
  RO7021594 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO7021594 - Day 10 |  |  |  |  |  |  |  | 7.85 (69.3) | 8.17 (100.8) | 10.7 (94.8) |
  RO7021594 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7021594 - Day 14 |  |  |  |  |  |  |  |  |  |  | 0.645 (44.2)
  RO7045755 - Day 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0
  RO7045755 - Day 1 | 1.17 (27.9) | 1.05 (36.2) | 0.918 (41.6) | 0.962 (19.8) | 1.03 (10.4) | 0.683 (53.1) | 0.744 (31.6) | 0.761 (36.0) | 0.657 (46.4) | 0.523 (37.9) |
  RO7045755 - Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7045755 - Day 3 |  |  |  |  |  |  |  |  |  |  | 0.612 (40.0)
  RO7045755 - Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 0
  RO7045755 - Day 10 |  |  |  |  |  |  |  | 0.744 (40.0) | 0.681 (52.4) | 0.536 (44.1) |
  RO7045755 - Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16
  RO7045755 - Day 14 |  |  |  |  |  |  |  |  |  |  | 0.645 (44.2)

24. Secondary Outcome: Part 3: Tmax of Midazolam
Description: A single IV dose of 100 ug midazolam was administered on Day 1 and Day 13. A single oral dose 300 ug of midazolam was administered on Day 2 and Day 14. RO6953958 was administrated once daily at 210 mg from Day 3 up to Day 14 so concomitantly with IV dose of midazolam on Day 13 and with oral dose of midazolam on Day 14.
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
Hour (h)
  Day 1 | 0.08 [0.08 to 0.08]
  Day 2 | 0.75 [0.50 to 1.50]
  Day 13 | 0.08 [0.08 to 0.25]
  Day 14 | 0.63 [0.50 to 1.00]

25. Secondary Outcome: Part 3: Cmax of Midazolam
Description: as for outcome 24
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
ng/mL
  Day 1 | 2410 (22.8)
  Day 2 | 1200 (28.5)
  Day 13 | 2030 (24.1)
  Day 14 | 1250 (31.2)

26. Secondary Outcome: Part 3: T1/2 of Midazolam
Description: as for outcome 24
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
h
  Day 1 | 4.38 (30.0)
  Day 2 | 4.44 (27.2)
  Day 13 | 4.69 (33.8)
  Day 14 | 4.55 (26.6)

27. Secondary Outcome: Part 3: AUClast of Midazolam
Description: as for outcome 24
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
h*ng/mL
  Day 1 | 3550 (22.8)
  Day 2 | 4140 (37.4)
  Day 13 | 3790 (25.8)
  Day 14 | 4470 (46.0)

28. Secondary Outcome: Part 3: AUCinf of Midazolam
Description: as for outcome 24
Time Frame: Day 1-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
h*ng/mL
  Day 1 | 3630 (24.4)
  Day 2 | 4270 (39.9)
  Day 13 | 3910 (29.2)
  Day 14 | 4630 (49.6)

29. Secondary Outcome: Part 3: VF of Oral Midazolam
Time Frame: Day 2-14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
Litre (L)
  Day 2 | 450 (32.0)
  Day 14 | 426 (32.1)

30. Secondary Outcome: Part 3: RAUC of Midazolam
Time Frame: Days 13 and 14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
Ratio
  Day 13 | 1.07 (10.3)
  Day 14 | 1.08 (20.7)

31. Secondary Outcome: Part 3: RCmax of Midazolam
Time Frame: Days 13 and 14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
Ratio
  Day 13 | 0.844 (22.8)
  Day 14 | 1.05 (22.5)

32. Secondary Outcome: Part 3: CL: Total Plasma Clearance of IV Midazolam
Time Frame: Days 1 and 13
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
L/h
  Day 1 | 27.6 (24.4)
  Day 13 | 25.6 (29.2)

33. Secondary Outcome: Part 3: Fraction Absorbed (F) of Midazolam
Description: F is stated as a fraction of 1.
Time Frame: Days 2 and 14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
Ratio
  Day 2 | 0.391 (22.0)
  Day 14 | 0.396 (23.9)

34. Secondary Outcome: Part 3: Volume of Distribution Under Steady-state Conditions (Vss) of Midazolam
Time Frame: Days 3 and 14
Population: The PK population included all participants who received active (RO6953958) treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
Number analyzed (Participants) | 16
Liters
  Day 3 | 161 (58.3)
  Day 14 | 142 (72.5)

ADVERSE EVENTS:
Time Frame: Part 1: From randomization up to 7 weeks (or up to 14 weeks if the participant is part of the food effect cohort). Parts 2 and 3: From randomization up to 8 weeks
Arm/Group | Part 1 (SAD): RO6953958 5mg (Fasted) | Part 1 (SAD): RO6953958 15mg (Fasted) | Part 1 (SAD): RO6953958 45mg (Fasted) | Part 1 (SAD): RO6953958 90mg (Fasted or Fed) | Part 1 (SAD): RO6953958 180mg (Fasted) | Part 1 (SAD): RO6953958 360mg (Fasted) | Part 1 (SAD): Placebo (Fasted) | Part 1 (SAD): Placebo (Fed) | Part 2 (MAD): RO6953958 45mg | Part 2 (MAD): RO6953958 140mg | Part 2 (MAD): RO6953958 210mg | Part 2 (MAD): Placebo | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 2/6 | 4/6 | 2/6 | 3/6 | 2/10 | 0/2 | 4/6 | 6/6 | 4/6 | 2/6 | 10/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (SAD): RO6953958 5mg (Fasted) (N=6) | Part 1 (SAD): RO6953958 15mg (Fasted) (N=6) | Part 1 (SAD): RO6953958 45mg (Fasted) (N=6) | Part 1 (SAD): RO6953958 90mg (Fasted or Fed) (N=6) | Part 1 (SAD): RO6953958 180mg (Fasted) (N=6) | Part 1 (SAD): RO6953958 360mg (Fasted) (N=6) | Part 1 (SAD): Placebo (Fasted) (N=10) | Part 1 (SAD): Placebo (Fed) (N=2) | Part 2 (MAD): RO6953958 45mg (N=6) | Part 2 (MAD): RO6953958 140mg (N=6) | Part 2 (MAD): RO6953958 210mg (N=6) | Part 2 (MAD): Placebo (N=6) | Part 3 (DDI): RO6953958 210mg, Midazolam Injection 100ug, Midazolam Oral 330ug (N=16)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Catheter Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter Site Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Medical Device Site Dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Puncture Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Procedural Headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness Postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | NA | 2 (2) | 3 (4) | 2 (3) | 1 (2) | 7 (7)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT04475848/Prot_SAP_000.pdf